CLINICAL TRIAL: NCT04405206
Title: Total Neoadjuvant Therapy Followed by 'Watch and Wait' Approach or Organ Preservation for MRI Stratified Low-risk Rectal Cancer: a Multi-center, Prospective, Single-arm Phase II Trial.
Brief Title: Total Neoadjuvant Therapy Followed by 'Watch and Wait' Approach or Organ Preservation for Low-risk Rectal Cancer
Acronym: BJCC-R01
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Aiwen Wu, Professor, Peking University Cancer Hospital & Institute
Other Study IDs: BJCC-R01
Record Dates: First submitted 2020-05-23; First posted 2020-05-28 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Rectum Cancer
Keywords: rectum cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Capecitabine; Radiotherapy, Intensity-Modulated; Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — FFPE and peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A:Clinical complete response (cCR): Group A:Clinical complete response (cCR) Patients who achieve cCR when restaged by DRE-Endoscopy-MRI-CEA at 16 weeks following intensity modulated radiotherapy(IMRT) plus consolidation CapeOX(Capecitabine+Oxaliplatin) will receive Nonoperative Management(NOM).
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Radiation: intensity modulated radiotherapy; Procedure: DRE-Endoscopy-MRI-CEA; Procedure: Nonoperative Management; Behavioral: Quality of Life Questionnaires
- Group B:Near-cCR: Patients who achieve near-cCR when restaged by DRE-Endoscopy-MRI-CEA at 16 weeks following intensity modulated radiotherapy(IMRT) plus consolidation CapeOX(Capecitabine+Oxaliplatin) will receive Local Excision(LE) or Nonoperative Management(NOM).
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Radiation: intensity modulated radiotherapy; Procedure: DRE-Endoscopy-MRI-CEA; Procedure: Nonoperative Management; Procedure: Local excision; Behavioral: Quality of Life Questionnaires
- Group C:Residual tumor: Patients with residual tumor when restaged by DRE-Endoscopy-MRI-CEA at 16 weeks following intensity modulated radiotherapy(IMRT) plus consolidation
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Radiation: intensity modulated radiotherapy; Procedure: DRE-Endoscopy-MRI-CEA; Procedure: Total Mesorectal Excision; Behavioral: Quality of Life Questionnaires

INTERVENTIONS:
Drug: Oxaliplatin — OXA 130mg/m2
  Other Names: OXA
Drug: Capecitabine — Cape 1000mg/m2
  Other Names: Cape
Radiation: intensity modulated radiotherapy — IMRT 50.4Gy/22f
  Other Names: IMRT
Procedure: DRE-Endoscopy-MRI-CEA — examination process in follow up
Procedure: Nonoperative Management — Watch and Wait
  Other Names: NOM
  Groups: Group A:Clinical complete response (cCR); Group B:Near-cCR
Procedure: Local excision — For ymriT1N0 and near-cCR patients，LE is optional.
  Other Names: LE
  Groups: Group B:Near-cCR
Procedure: Total Mesorectal Excision — Standard TME surgery openly or laporoscopically
  Other Names: TME
  Groups: Group C:Residual tumor
Behavioral: Quality of Life Questionnaires — QLQ C30 and QLQ CR29
  Other Names: QLQ

SUMMARY:
Aim: To investigate the safety and efficacy of organ preservation (OP) with watch-and-wait strategy (W&W) or local excision (LE) in MRI stratified low-risk rectal cancer treated by total neoadjuvant treatment. Meanwhile we will look into the role of ctDNA in the prediction of regrowth and metastasis in the wait and wait process.

Methods: Low-risk rectal cancer with following MRI features are recruited: mid-low tumor, mrT2-3b, MRF(-), EMVI(-), differentiation grade 1-3. Patients will receive IMRT 50.6Gy/22f with concurrent capecitabine and 4 cycles of consolidation CAPEOX. Patients with cCR/near-cCR were recommended for 'watch & wait' approach or local excision (LE). The OPR and sphincter preservation rate (SPR) at 2 years will be analyzed.

As the extension of PKUCH-R01, BJCC-R01 trial will upgrade to a multi-center research enrolled 3 other colorectal center in Beijing.

DETAILED DESCRIPTION:
Neoadjuvant chemoradiotherapy (nCRT), total mesorectal excision and adjuvant chemotherapy comprise the standard treatment for locally advanced rectal cancer, following which 15-30% patients achieved pathological complete response need to receive the removal of rectum without residual tumor and suffer significant functional impairment even after sphincter preservation. Adjuvant chemotherapy is also questioned for its benefit for prolonged survival through the data from various studies. More evidence demonstrated that organ-preservation (e.g. non-operative management or local excision) for patients with clinical complete response (cCR) or near-cCR following nCRT had similar survival when compared with those received standard care.

This study is designed to investigate the efficacy of neoadjuvant intensity modulated nCRT with concurrent capecitabine plus consolidation CapeOX for T2/DWI/Enhanced MRI defined cT2-T3b mid-low rectal cancer without threatening mesorectal fascia or extramural vascular invasion (EMVI) or mrN2 disease.

According to the response to treatment evaluated by multi-modal assessment including digital exam, T2/DWI/Enhanced MRI, endoscopy and serum CEA test, patients will receive tailored operative management like local excision or total mesorectal excision, or non-operative management. Intention to treatment was also allowed in this study.

Firstly, the investigators will observe the organ preservation rate at 2 years. Endpoints for organ-preservation like non-regrowth DFS, stoma-free survival and other conventional survival outcomes (DFS, OS) would be further collected. The short-term and long-term QoL will be measured in all patients.

. Our baseline data showed the 48% of locally advanced rectal cancers could be downstaged to stage ypT0-2N0 following IMRT with concurrent capecitabine. We hypothesize that at least 24% of rectal cancers could be candidates for LE or NOM after IMRT and the rectum preservation rate will increase to 40% in low-risk rectal cancers by LE or NOM following IMRT plus consolidation CapeOX at 2 years. As a superiority design, this study need to recruit 64 patients to test this hypothesis, with 85% power (exact binomial test for proportions, alpha = 5 %, one-sided), If the number of responses is 22 or more, the hypothesis that P <= 0.240 is rejected. We anticipate about 10 % loss to follow-up, so we will recruit an additional 8 patients and the study will recruit 72 patients in all.

ELIGIBILITY:
Inclusion Criteria:

* 1. the age is more than 18 years old and less than 85 years old;
* 2. ECOG score of physical condition is 0-1;
* 3. adenocarcinoma of rectum confirmed by pathology; differentiated into Grade 1-3, i.e. high, medium and low differentiated adenocarcinoma
* 4. the distance from the lower edge of the tumor to the anal edge ≤ 12cm (endoscopy) or to the anorectal ring (ARJ) ≤ 8cm;
* 5. the initial MRI was T2 / T3a / T3B, with negative EMVI and negative CRM. There was no lymph node metastasis outside the ilium, general ilium, obturator and abdominal aorta
* 6. the maximum diameter of tumor ≤ 4cm or the circumferentially invasive area is less than 1 / 3 of intestinal circumference
* 7. no evidence of distant metastasis;
* 8. no history of pelvic radiotherapy;
* 9. no history of surgery or chemotherapy for rectal cancer;
* 10. systemic infection without antibiotic treatment;
* 11. blood routine test: neutrophil absolute value > 1.5 × 10 9 / L, HGB > 10.0 g / dl, PLT > 100 × 10 9 / L;
* 12. blood biochemistry: total bilirubin ≤ 1.5 x ULN, AST ≤ 3 x ULN, ALT ≤ 4 x ULN;
* 13. the patient read and signed the informed consent of the study and agreed to participate in the study;

Exclusion Criteria:

* 1. recurrent rectal cancer;
* 2. initial local non resectable rectal cancer (no possibility of R0 whole block resection);
* 3. the creatinine level is 1.5 times higher than the upper limit of normal value;
* 4. have a history of pelvic radiotherapy;
* 5. the patients could not tolerate the enhanced MRI;
* 6. malignant tumors whose survival rate in the past 5 years is significantly lower than that of rectal cancer in our center (excluding well treated basal cell carcinoma, skin squamous carcinoma, small renal carcinoma, breast cancer and thyroid papillary carcinoma);
* 7. in the past 6 months, the patients had arterial embolism diseases, such as angina, MI, TIA, CVA, etc;
* 8. have received other types of anti-tumor or experimental treatment;
* 9. the patients are pregnant or lactating women;
* 10. patients with other diseases or mental disorders may affect their participation in this study;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rectal cancer patient who receives primary care in Beijing Cancer Hospital will be selected as the candidate for this study.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2020-05-25 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
OPR(organ preservation rate) | 3 year
  Proportion of patients who achieved cCR or near cCR after neoadjuvant treatment and received watch and wait approach or local excision

SECONDARY OUTCOMES:
NR-DFS(Non-regrowth disease free survival) | 3 year
  Within 3 years after receiving the neoadjuvant treatment, the time patient in status free of death, local recurrence after radical resection or distant metastasis.
SFS(stoma-free survival) | 3 year
  Within 3 years after receiving the neoadjuvant treatment, the time patient in status free of stoma

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided